CLINICAL TRIAL: NCT01568346
Title: Randomized Trail of Breast MRI for Newly Diagnosed Early Stage Breast Cancer: Impact on Re-excision Lumpectomy
Brief Title: Breast MRI for Newly Diagnosed Breast Cancer:Impact on Re-excision Lumpectomy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow Accural
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Mehra Golshan, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 11-330
Record Dates: First submitted 2012-03-29; First posted 2012-04-02 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-08

CONDITIONS: Breast Cancer
Keywords: Newly diagnosed; Early stage
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MRI (Active Comparator): MRI
  Interventions: Other: MRI
- No MRI (No Intervention): No MRI

INTERVENTIONS:
Other: MRI — Breast MRI
  Arms: MRI

SUMMARY:
This study is being done to find out the number of surgical procedures required to achieve clear margins in women with newly diagnosed early stage breast carcinoma. The investigators are also looking at the number of additional biopsies performed before surgery, the mastectomy rate, detection of breast cancer on the opposite side (contralateral carcinoma), time form diagnosis to local therapy, and evaluation time to local recurrence.

DETAILED DESCRIPTION:
This is a prospective pragmatic trial randomizing women diagnosed with early stage breast cancer to MRI versus no breast MRI. Data analyzed will include medical record information abstracted from the clinical records. Date and modality of all imaging performed, malignancy(s) identified, abnormalities identified, image guided procedures performed, surgical procedures performed and pathology results.

The primary aim of this study is to assess if the use of pre-operative MRI can reduce the incidence of re-excisions required to achieve clear margins in women with newly diagnosed early stage breast carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Must undergo definitive local therapy with either breast conserving therapy or mastectomy
* Clinical Stage 0, I or II breast cancer based on examination and/or conventional imaging of mammogram with or without ultrasound. Tumors must be less than 5 cm in size and the patient clinically node negative
* Able to undergo breast MRI

Exclusion Criteria:

* Not pregnant or breastfeeding
* No prior breast MRI for the newly diagnosed carcinoma at the outside hospital
* No prior mantle radiation
* No locally advanced breast cancer
* No diffuse malignant appearing microcalcifications requiring mastectomy
* No known collagen vascular disease
* No previous ipsilateral radiation
* No participants who undergo surgery at an outside institution
* No prior history of breast carcinoma

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Assess if pre-operative MRI reduces incidence of re-excisions required | 2 years
  Assess if the use of pre-operative MRI can reduce the incidence of re-excisions required to achieve clear margins in women with newly diagnosed early stage breast carcinoma

SECONDARY OUTCOMES:
Total Mastectomy Rates | 2 years
  Total Mastectomy Rates
Number of biopsies | 2 years
  The number of biopsies recommended and performed
Local-regional recurrence rates | 2 years
  Local-regional recurrence rates in participants undergoing local therapy
Time from diagnosis to local therapy | 2 years
  The time from diagnosis to definitive local therapy
Number of malignancies in contralateral breast | 2 years
  The number of malignancies identified int he contralateral breast

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Faulkner Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No